CLINICAL TRIAL: NCT03871465
Title: Effect of Combined Ultrasound-guided Subdeltoid Corticosteroid Injections and Physiotherapy in Treatment of Patients With Chronic Subacromial Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20171205R; NSTC 107-2314-B-341-002 (Other Grant/Funding Number: National Science and Technology Council); NSTC 108-2314-B-341-002 (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2018-09-06; First posted 2019-03-12 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Subacromial Bursitis; Subacromial Impingement Syndrome; Physical Therapy; Therapeutic Exercise; Rehabilitation
Keywords: subacromial bursitis; subacromial impingement syndrome; corticosteroid; physical therapy; therapeutic exercise; rehabilitation
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triamcinolone SASD injection (Experimental): 2ml triamcinolone (1ml/10mg) and 3ml 1% xylocain will be injected into the affected SASD bursa under ultrasound guidance.
  Interventions: Drug: Triamcinolone SASD injection
- Physiotherapy (Experimental): The physiotherapy program consists of hot pack, interferential therapy, and exercise program, which includes stretch exercise, mobilization of the glenohumeral joint, manual pressure to the possible trigger points, scapular stabilization exercise, and strengthening exercise of the rotator cuff, trapezius, and serratus anterior muscles.
  Interventions: Procedure: Physiotherapy
- Triamcinolone injections & Physiotherapy (Experimental): 2ml triamcinolone (1ml/10mg) and 3ml 1% xylocain will be injected into the affected SASD bursa under ultrasound guidance.
  The physiotherapy program consists of hot pack, interferential therapy, and exercise program, which includes stretch exercise, mobilization of the glenohumeral joint, manual pressure to the possible trigger points, scapular stabilization exercise, and strengthening exercise of the rotator cuff, trapezius, and serratus anterior muscles.
  Interventions: Drug: Triamcinolone injections & Physiotherapy

INTERVENTIONS:
Drug: Triamcinolone SASD injection — 2ml triamcinolone (1ml/10mg) and 3ml 1% xylocain will be injected into the affected SASD bursa under ultrasound guidance.
  Arms: Triamcinolone SASD injection
Procedure: Physiotherapy — The physiotherapy program consists of hot pack, interferential therapy, and exercise program, which includes stretch exercise, mobilization of the glenohumeral joint, manual pressure to the possible trigger points, scapular stabilization exercise, and strengthening exercise of the rotator cuff, trapezius, and serratus anterior muscles.
  Arms: Physiotherapy
Drug: Triamcinolone injections & Physiotherapy — 2ml triamcinolone (1ml/10mg) and 3ml 1% xylocain will be injected into the affected SASD bursa under ultrasound guidance.
  The physiotherapy program consists of hot pack, interferential therapy, and exercise program, which includes stretch exercise, mobilization of the glenohumeral joint, manual pressure to the possible trigger points, scapular stabilization exercise, and strengthening exercise of the rotator cuff, trapezius, and serratus anterior muscles.
  Arms: Triamcinolone injections & Physiotherapy

SUMMARY:
This study is to investigate whether combination of ultrasound-guided subdeltoidcorticosteroid injection and physiotherapy is more effective than either treatment alone in treatment of patients with chronic subacromial (or subdeltoid) bursitis (SAB).

DETAILED DESCRIPTION:
Chronic subacromial bursitis (SAB) is a common shoulder disorder characterized by chronic shoulder pain with a painful arc of motion, and/or pain on active or passive motions. The diagnosis of SAB requires confirmation by an infiltration with local anesthetic. Previous study showed that corticosteroid injection is more effective than hyaluronic acid in treatment of chronic SAB, however, some (about 20%) patients were not responsive to corticosteroid injection, and some responsive patients may have recurrence of symptoms. The purpose of this study is to investigate whether combination of corticosteroids SASD injections and physiotherapy is more effective than either treatment alone in chronic SAB.

ELIGIBILITY:
Inclusion Criteria:

1. shoulder pain for more than 1 month
2. age ≥20 years old
3. painful abduction or internal rotation with a visual analog scale (VAS) pain score ≥4
4. the presence of a painful arc of motion or pain at the middle to terminal range of shoulder abduction or internal rotation with an empty or soft end feel
5. positive shoulder impingement test (Neer test and/or Hawkin test)
6. a reduction in pain of ≥40% on active shoulder abduction or internal rotation at the terminal range after injection of 3ml of 1%lidocain into the SASD bursa under US guidance.

Exclusion Criteria:

1. a history of uncontrolled chronic diseases, e.g., malignant neoplasms, blood dyscrasia, and serious infection
2. previous surgery of the affected shoulder
3. any evidence of a rotator cuff tear or tendinopathy, demonstrated by positive resistive tests andsonographic findings
4. calcification of the rotator cuff, demonstrated by x-ray or sonographic findings
5. the presence of arthritis, such asinflammatory arthritis(e.g., rheumatoid arthritis, seronegativespondyloarthropathy, or crystal-related arthropathy), osteoarthritis, frozen shoulder, subacromial spurs, or deformity of the acromion
6. the presence of instability of the affected shoulder
7. a previous fracture near the shoulder region
8. the presence of cervical radiculopathy or myelopathy
9. having received a corticosteroid or hyaluronic acid subacromial or shoulder joint injection in the past 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
The pain VAS score | change between baseline and at 8 weeks after the beginning of the treatment.
  The pain VAS score is obtained using a 100-mm-long horizontal line, with 0 mm on the left indicating no pain and 100 mm on the right indicating very severe pain.
The scores of the Shoulder Pain and Disability Index (SPADI) | change between baseline and at 8 weeks after the beginning of the treatment.
  The total SPADI score, which ranges between 0 and 100, is calculated by averaging the scores from the pain and disabilities subclasses.

SECONDARY OUTCOMES:
The active ROM | change between baseline and at 8 weeks after the beginning of the treatment.
  The maximal active ROMs of the affected shoulder will be measured using a goniometer under the guidelines of the American Academy of Orthopedic Surgeons. These measurements included abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0 degrees of abduction.
Change of the Shoulder Disability Questionnaire (SDQ) | change between baseline and at 8 weeks after the beginning of the treatment.
  The SDQ is a symptoms-related questionnaire containing 16 items describing common situations that may induce symptoms in patients with shoulder disorders. By responding 'yes', 'no', or 'not applicable', the final score is obtained by dividing the number of positively scored items by the total number of applicable items and then multiplying this number by 100, which results in a final score ranging between 0 (no disability) and 100 (the worst situation).
The Western Ontario Rotator Cuff Index (WORC). | change between baseline and at 8 weeks after the beginning of the treatment.
  It is composed of 5 subscales: physical symptoms, sports/recreation, work, lifestyle, and emotions. Each item has a score range of 0 to 100.Scores can be computed for individual subscales and summated for a total score, which can range from 0-2100, with a higher score representing lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan